CLINICAL TRIAL: NCT03808675
Title: Long Term Aerobic Exercise to Slow Progression in Parkinson's Disease
Brief Title: Aerobic Exercise in Parkinson's Disease
Acronym: LTAE-PD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E2987-R; 1I01RX002987-01A1 (NIH)
Record Dates: First submitted 2019-01-07; First posted 2019-01-17 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Exercise; Aerobic exercise; Cognition; Driving; Diffusion tensor imaging; DTI; MRI; Depression; Cardiorespiratory Fitness; Quality of life; Health education; Executive functions
MeSH Terms: conditions — Parkinson Disease; Motor Activity; Depression; Health Education

STUDY DESIGN:
Intervention Model Description: One-year, single-blind, parallel group, randomized controlled trial (RCT) that compares the effects of moderate aerobic exercise vs. usual care + health education
Who Masked: Outcomes Assessor
Masking Description: Due to nature of the intervention (exercise), the participant cannot be blinded. However, assessors for various outcomes will be blinded to the group status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aerobic (Experimental): Participants randomized to aerobic exercise
  Interventions: Behavioral: Aerobic walking
- Control (Other): Participants randomized to usual care with PD specific health education
  Interventions: Behavioral: Usual care with PD specific health education

INTERVENTIONS:
Behavioral: Aerobic walking — The investigators will use self-administered continuous walking exercise at a moderate intensity level, defined as 40-59% of heart rate reserve or 64-77% of heart rate at gas exchange threshold (HRGET) by ACSM as in the investigators' preliminary study (PMID: 24991037 PMCID: PMC4132568). The HRGET will be determined as the heart rate at VO2max during graded cycle ergometry. The total duration of the exercises will be 150 min/week per 2008 Physical Activity Guidelines for Americans and American Heart Association recommendations, conducted in three 50 min sessions. The aerobic walking intervention will take place outdoors (e.g., trails, sidewalks, parks) or indoors (e.g., track in a local gym or a mall) depending on the preferences of the subject and weather. Session duration will be 20 min the first week and will be advanced by 5 min per week over 6 weeks.
  Arms: Aerobic
Behavioral: Usual care with PD specific health education — In this study, patients will receive their usual medical treatment for motor and non-motor symptoms from their
  primary neurologist. The investigators will use a streamlined form of PD specific health education prepared by the VA: My Parkinson's Story, which consists of a series of short videos prepared by the VA PADRECCs addressing various aspects of PD. These 6-12 minutes long videos are freely available on YouTube. The investigators can also provide them on a CD if subjects desire. They start with a patient testimony about the topic of the episode, followed by comments of experts in the field. The title of the episodes are: Early Parkinson's, Medications, Exercise, Memory, Visual Disturbances, Depression, Sleep, Speech and Swallowing, Impulsive Behaviors, Driving, Pain, Dyskinesias, Deep Brain Stimulation, Advanced Parkinson's Disease, Falls, The Caregiver, Hospitalization, Genetics, Environmental Exposure, Atypical Parkinsonism
  Arms: Control

SUMMARY:
Parkinson's disease (PD) is an incurable brain illness that afflicts more than one million Americans, including many aging Veterans. PD places an unbearable burden on the individual due to progressive impairment of movement and mental function. As a result, patients lose critical abilities such as driving and can become isolated. Although drugs and surgery help movement problems, their benefits are temporary and may cause side effects. Drugs provide limited and temporary benefit for cognition and do not prevent dementia. Animal and preliminary human studies on aerobic exercise show promising results in helping a broad spectrum of symptoms. However, due to limited and inconsistent research results, the long term effects of aerobic exercise on brain health and clinical features in PD is unknown. The investigators will conduct a clinical trial to test the long term effects of aerobic exercise on the brain tissue, movement, mental functions, and driving in PD. If effective, aerobic exercise can be implemented immediately as a low cost, easily accessible treatment in PD.

DETAILED DESCRIPTION:
Parkinson's disease (PD) culminates in dementia, immobility, and death at a huge societal cost. Even early in the course, motor and cognitive dysfunction impairs instrumental activities of daily living (IADL). Non-motor symptoms due to fatigue, mood, sleep, and autonomic disorders further reduce quality of life (QoL). DTI shows progressive decline in brain tissue integrity. Usual care of PD centers on medical and surgical treatments relieve motor symptoms, but these cause side effects and lose efficacy over time. Usual treatment for non motor manifestations with pharmaceuticals (e.g., antidepressants) is symptomatic and not specific for PD. Acetylcholine esterase inhibitors exert modest symptomatic benefits on dementia, but there is no approved treatment for mild cognitive impairment. Physical Therapy is usually prescribed in later stages when mobility impairment ensues. There is no approved standard exercise regimen for PD. There is no cure or disease modifying treatment. Thus, there is a critical need for treatments that provide broad spectrum of benefits and slow PD.

Preliminary research suggests that aerobic exercise has potential to meet this need. However, aerobic exercise is demanding and carries some risks. It is unknown if aerobic exercise is more beneficial than usual care in PD in long term due to gaps in the investigators knowledge about the effects of cardiorespiratory fitness (CRF) on brain tissue integrity, motor function, cognition, IADL, QoL, and disease progression. Limitations of current studies include short duration, small sample size, lack or inadequacy of controls, lack of outcome measures for cognition and IADL, and lack of biological markers to measure progression. The objective in this application is to fill the translational gap by determining the biological, clinical, and functional effects of long term aerobic exercise (LTAE) in PD.

The overall hypothesis is that LTAE improves brain tissue integrity and slows down PD. The FIRST AIM is to determine the effects of LTAE on clinical features and functional abilities in PD. The investigators' prior 6-month, uncontrolled trial showed preliminary evidence that aerobic exercise improves aspects of motor function, cognition, and QoL in PD, but long term outcomes and implication for functional abilities are unknown. The investigators hypothesize that LTAE will provide sustained improvement in motor function, cognition, and non-motor symptoms with translation of benefits to QoL and IADL. The investigators will test this with a one-year randomized controlled trial (RCT) that compares the effects of moderate aerobic exercise vs usual care. The investigators will use driving as the outcome for IADL. Driving represents an important symbol for independence, and depends on integrity of cognitive and motor systems. The SECOND AIM is to determine the mechanism of LTAE effects in PD. CRF reflects complex improvements in vascular, cardiac, and metabolic health from aerobic exercise. There is preliminary evidence that higher CRF is associated with better brain health and motor/cognitive function, and that aerobic exercise improves these outcomes. For example, the investigators' preliminary study showed improvement of microtissue integrity in the striatum and white matter on DTI, but it is unclear how these changes counteract PD progression over long term. The hypotheses are: 1) LTAE will improve brain tissue integrity as indexed by DTI, 2) LTAE effects on motor and cognitive function are mediated by changes in brain tissue integrity on DTI, and 3) physiological processes leading to improved CRF from AE are critical to the benefits on the brain tissue integrity and motor/cognitive function. The investigators will test these hypotheses determining the effects of LTAE on CRF and DTI, and the association between individual differences in training related changes in motor and cognitive function, DTI, and CRF.

In summary, the investigators' proposal leverages the diverse interdisciplinary team, strong preliminary data and past work, and unique infrastructure to determine if LTAE slows down neurodegeneration and clinical disability in PD.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 40 and older with the diagnosis of idiopathic PD per UK Brain Bank criteria
* Hoehn-Yahr Stage I-III, on stable dopaminergic treatment regimen for equal or greater than 4 weeks prior to baseline.
* Aerobic Fitness: VO2max below "very good" fitness levels for their age and gender at baseline cyle ergometry.

To include subjects who have room to improve their aerobic fitness, the investigators will enroll only those subjects whose VO2max is below "very good" fitness level (about 90% of the population) using age and gender based VO2max norms based review of 62 studies where VO2max was measured directly in healthy adult subjects in the USA, Canada and 7 European countries (Reference: Shvartz, E and Reibold, RC. Aerobic fitness norms for males and females aged 6 to 75 years: a review.

Aviat Space Environ Med. 1990; 61:3-11).

* Cognitive function: No dementia per Movement Disorder Society Level I criteria (Reference: Dubois, B, Burn, D, Goetz, C, et al. Diagnostic procedures for Parkinson's disease dementia: recommendations from the movement disorder society task force. Mov Disord. 2007; 22:2314-2324).
* Current active drivers with a valid driver's license
* Veteran or non-veteran

Exclusion Criteria:

* Subjects unwilling or unable to give informed consent
* Secondary parkinsonism (e.g., drug induced)
* Parkinson-plus syndromes
* History of brain surgery for PD such as deep brain stimulation
* Corrected visual acuity less than 20/50 (due to effect on driving)
* Contraindications to exercise per ACSM criteria for Exercise Testing and Training (Reference: American College of Sports Medicine. Cardiorespiratory Exercise Prescription. In: Ehrman JK, ed. ACSM's Guidelines for Exercise Testing and Prescription.6th ed. Baltimore: Lippincott Williams & Wilkins, 2010:448-462).
* No confounding acute or unstable medical, psychiatric, orthopedic condition. Subjects who have hypertension, diabetes mellitus, depression, or other common age related illness will be included if their disease under control with stable treatment regimen for at least 30 days.
* Clinically significant TBI or PTSD
* Presence of other known medical or psychiatric comorbidity that in the investigator's opinion would compromise participation in the study
* Presence of dementia per Movement Disorder Society Level I criteria
* Subjects with clinically significant depression as determined by a Beck Depression Inventory (BDI) score greater than 15 at the screening visit
* History of exposure to typical or atypical antipsychotics or other dopamine blocking agents within 6 months prior to the baseline visit
* Use of investigational drugs within 30 days before screening
* Subjects have to be on a stable regimen of central nervous system acting medications (benzodiazepines, antidepressants, hypnotics) for 30 days prior to the baseline visit
* Contraindication to having a brain MRI

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
OFF period MDS-UPDRS Motor Subscale score | Change from Baseline OFF period MDS-UPDRS Motor Subscale score at 1 year
  Motor function. MDS-UPDRS motor examination subscale (Part III) score in the "practically defined OFF state", i.e., after overnight (~12 hours) withdrawal of PD medications. Higher scores worse. Range: 0-132.
Percent Increase Score (PIS) on Eriksen's flanker task | Change from Baseline Percent Increase Score (PIS) on Eriksen's flanker task at 1 year
  Cognitive function. Due to its sensitivity to changes in aerobic fitness (including in the investigators' preliminary study), the investigators chose change in Percent Increase Score (PIS) on Eriksen's flanker task, which measures the cost of conflict resolution between the incongruent and congruent stimuli. Higher scores worse.
total number of driving safety errors on road test | Change from Baseline total number of driving safety errors on road test at 1 year
  Driving. The video of a standardized experimental drive in an instrumented vehicle will be scored for safety errors by a certified driving instructor. Higher scores worse.
regional DTI (diffusion tensor imaging) | Change from Baseline regional DTI at 1 year
  Brain tissue integrity. The investigators will analyze differences in regional rD (radial diffusivity) changes between the aerobic exercise and usual care control groups in primary outcome regions of interest (Putamen, Cingulum, Superior Longitudinal Fasciculus). Higher scores worse.
MDS-UPDRS Non-motor Experiences of Daily Living subscale (Part I) score | Change from Baseline MDS-UPDRS Non-motor Experiences of Daily Living subscale (Part I) score at 1 year
  Non-motor symptoms. Higher scores worse. Range: 0-48
Summary index of the Parkinson's Disease Questionnaire-39 (PDQ-39) | Change from Baseline PDQ-39 Summary Index at 1 year
  Quality of life

SECONDARY OUTCOMES:
ON Period MDS-UPDRS motor examination subscale score | Change from Baseline ON Period MDS-UPDRS motor examination subscale score at 1 year
  Motor function. Higher scores worse. Range: 0-132.
Dexterity (time on 9-hole peg board) test of NIH Toolbox motor battery | Change from Baseline 9-hole peg board test performance at 1 year
  Motor function. Dexterity
COGSTAT score | Change from Baseline COGSTAT score at 1 year
  Cognitive function. COGSTAT, a composite measure of cognition, calculated by assigning and summing standard T-scores (mean=50, SD=10) to eight tests from the cognitive test battery the investigators used in the driving studies, will be the main secondary outcome measure. This cognitive battery will enable us to probe multiple domains: Complex Figure Test-Copy (CFT-Copy) Version, Block Design for visuospatial construction; Trail-making Test (B-A), a measure of set shifting and Controlled Oral Word Association Test (also tests language) for executive functions; Rey Auditory Verbal Learning Test (anterograde verbal memory), CFT-Recall is administered 30 minutes after the CFT-Copy (visual memory), Benton Visual Retention Test errors for memory; Judgment of Line Orientation for visual perception. Higher scores worse.
Radial Diffusivity (rD) on Diffusion imaging tractography | Change from Baseline Diffusion imaging tractography at 1 year
  Brain tissue integrity. Motor: Substantia nigra <-> putamen (nigrostriatal tract) and putamen <-> premotor cortex Cognitive: Dorsal lateral prefrontal cortex (DLPFC) <-> caudate and the parietal cortex <-> prefrontal cortex. Higher scores worse.
Geriatric Depression Scale (GDS) score | Change from Baseline GDS score at 1 year
  Severity of depression. Higher scores worse. Range: 0-15
Motor experiences of daily living score | Change from Baseline motor experiences of daily living score at 1 year
  Motor function. Higher scores worse. Range:0-52.
Beck Anxiety Inventory (BAI) score | Change from Baseline BAI score at 1 year
  Anxiety severity. Higher scores worse. Range: 0-63
Parkinson's Disease Sleep Scale version 2 (PDSS-2) | Change from Baseline PDSS-2 score at 1 year
  Sleep quality. Higher scores worse. Range: 0-60
Fatigue Severity Scale (FSS) | Change from Baseline FSS score at 1 year
  Severity of fatigue. Higher scores worse. Range: 9-63
Locomotion (time on 25-f walk test for gait speed) test | Change from Baseline Locomotion (time on 25-f walk test for gait speed) test performance at 1 year
  Motor function. Locomotion.
Locomotion (time on 4-m walk test for gait speed) test of NIH Toolbox motor battery | Change from Baseline Locomotion (time on 4-m walk test for gait speed) test performance at 1 year
  Motor function. Locomotion
Finger Tapping test | Change from Baseline average performance for right and left finger tapping at 1 year
  Average between two trials of oscillating finger tapping for both hands.
Endurance (distance on 6-minute walk) test | Change from Baseline Endurance (distance on 6-minute walk) test performance at 1 year
  Motor function. Endurance (6-minute walk).
Schwab and England Activities of Daily Living Scale | Change from Baseline score at 1 year
  Changes of ability to complete activities of daily living. Lower percentage of ability worse. Range: 0-100%
Mini-Mental Status Examination (MMSE) | Change from Baseline MMSE score at 1 year
  Cognitive and memory. Lower scores worse. Range: 0-30
Montreal Cognitive Assessment (MOCA) | Change from Baseline MOCA score at 1 year
  Cognitive and memory. Lower scores worse. Range: 0-30
Pelli-Robson Contrast Sensitivity | Change from Baseline score at 1 year
  Vision. Sensitivity to contrast changes of letters. Range: 0.00 - 2.25
Early Treatment Diabetic Retinopathy Study (ETDRS) | Change from Baseline score at 1 year
  Visual acuity test. Changes of ETDRS Acuity Log Score.
EEG | Change from Baseline metrics at 1 year
  Various EEG metrics.

OTHER OUTCOMES:
VO2max on cycle ergometry | Change from Baseline VO2max on cycle ergometry at 1 year
  Cardiorespiratory fitness as an index of aerobic exercise intervention delivery. Higher scores better.

CONTACTS AND LOCATIONS:
Overall Officials: Ergun Y. Uc, MD, Principal Investigator — Iowa City VA Health Care System, Iowa City, IA
Locations (2):
- United States (2):
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa

IPD SHARING:
Plan to Share IPD: Yes
Final datasets underlying all publications resulting from the proposed research will be shared outside VA.
  Final data sets underlying publications resulting from this research will be shared upon written request and through ClinicalTrials.gov and databank/repository if specified by the VA.
  Individuals can download the data and analyze the results using methods described in the investigators' articles or alternative methods as necessary.
Time Frame: As per VA specifications.
Access Criteria: As per VA specifications.

REFERENCES:
- [Background] Uc EY, Doerschug KC, Magnotta V, Dawson JD, Thomsen TR, Kline JN, Rizzo M, Newman SR, Mehta S, Grabowski TJ, Bruss J, Blanchette DR, Anderson SW, Voss MW, Kramer AF, Darling WG. Phase I/II randomized trial of aerobic exercise in Parkinson disease in a community setting. Neurology. 2014 Jul 29;83(5):413-25. doi: 10.1212/WNL.0000000000000644. Epub 2014 Jul 2. PMID 24991037

DOCUMENTS (1):
  • Informed Consent Form (2023-01-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT03808675/ICF_000.pdf